CLINICAL TRIAL: NCT00240071
Title: The Study of Avastin (Bevacizumab) to Reverse Acquired Estrogen Independence in Metastatic Breast Cancer Patients Previously Responsive to Hormonal Therapy: A Phase II Trial
Brief Title: Study of Avastin (Bevacizumab) to Reverse Acquired Estrogen Independence in Previously Hormone Responsive Metastatic Breast Ca.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Carla Falkson, MD, Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F050103001; UAB 0461 (Other: institutional protocol study number)
Record Dates: First submitted 2005-10-13; First posted 2005-10-17 (Estimated); Results first posted 2011-09-27 (Estimated); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Metastatic Breast Cancer
Keywords: Breast cancer; Metastatic breast cancer; Hormonal therapy; Bevacizumab
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab; Letrozole; Anastrozole; exemestane; Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Avastin (Experimental): The patient will continue the same hormonal therapy used prior to study enrollment but will combine it with Avastin.
  Interventions: Drug: Avastin; Drug: Hormonal therapy

INTERVENTIONS:
Drug: Avastin — All patients will received Avastin 15 mg/kg IV every three weeks. The first evaluation will be done at Week 6. Patients with objective response or stable disease will continue therapy with restaging every 6 weeks until evidence of disease progression. Patients with progression of disease will be taken off study.
  Other Names: Bevacizumab
Drug: Hormonal therapy — aromatase inhibitor (letrozole 2.5mg/d PO, anastrazole 1mg/d PO, or exemestane 25mg/d PO)or Selective Estrogen Receptor Modulator (SERM) (tamoxifen 20mg/d PO)
  Other Names: Femara (letrozole); Arimidex (anastrazole); Aromasin (exemestane); Nolvadex (tamoxifen)

SUMMARY:
The purpose of this study is to determine if acquired hormone therapy resistance can be reversed by Avastin (Bevacizumab), as measured by time to disease progression and evaluate toxicity of the combination of hormone treatment plus Avastin (Bevacizumab).

DETAILED DESCRIPTION:
This is a single institution, open-label study designed to evaluate safety and efficacy of Avastin (Bevacizumab) combined with an endocrine agent in patients with estrogen and/or progesterone receptor positive metastatic breast carcinoma who have acquired resistance to at least one hormonal agent. Patients will be treated with the same hormonal agent that was used previously assuming that the patient had a partial or complete response (for at least 6 months) followed by a clear disease progression using the Response Evaluation Criteria in solid Tumors (RECIST Criteria). Patients with stable disease for a prolonged time (for at least 6 months) will be also eligible to enter in the trial. Patients who have not had interval studies to evaluate disease response will be considered eligible if they have remained clinically stable (i.e. stable performance status (PS), no increasing pain) and on the same hormone for at least 6 months, and now they have signs and symptoms of clinical progression (i.e. elevated tumor markers, increasing bone pain, worsening performance status). Patients must have histologically confirmed measurable and/or evaluable metastatic breast cancer with positive estrogen and/or progesterone receptors. Patients can have up to an 8-12 week break in therapy (discontinuation of hormonal therapy) and still remain eligible for the study as long as the documentation of disease progression is determined before the 8-12 week break in hormonal therapy.

The type and dose of the hormonal agent that will be used in this trial will be the same one that the patient used before progression. Hormonal therapy may include any estrogen deprivation reagent such as Tamoxifen, Anastrazole, Exemestane, Letrozole, or Fulvestrant. All patients will receive Avastin (Bevacizumab) 15 mg/kg IV every three weeks. Based on statistical evaluations, 30 patients will be enrolled. The first evaluation of efficacy will be done at week 6; patients with objective response or stable disease will continue therapy with re-staging every 6 weeks until evidence of disease progression. Patients with progression of disease will be taken off study (see appendix A). PET scan will be done at baseline and only in the first evaluation (6 weeks) to obtain early "metabolic response data" that will be correlated with objective response and time to disease progression (PET data on week 6 will not be used to evaluate response and to make therapeutic decisions). PET "metabolic response" will be defined as a >20% reduction in Standardized Uptake Value (SUV). Safety will be assessed by the recording of adverse events, serious adverse events, laboratory test results, and changes in vital signs. A positive response to Avastin (Bevacizumab) (reversal of hormonal resistance) will be defined as an objective response or stable disease of ≥ 3 months duration. All concomitant medication must be documented. Additionally, any diagnostic, therapeutic or surgical procedure performed during the study period, should be recorded including the date, indication, description of the procedure(s) and any clinical findings.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have cytologically or histologically proven breast cancer which is estrogen receptor or progesterone receptor positive and is locally advanced and /or metastatic.
* Give written informed consent prior to study specific screening procedures, with the understanding that the patient has the right to withdraw from the study at any time, without prejudice (Appendix E).
* Be female and greater than or equal to 19 years of age (age limit required by the State of Alabama). Women of childbearing potential must have a negative pregnancy test and must be willing to consent to using effective contraception while on treatment and for a reasonable period thereafter. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Be ambulatory (outpatient) and have an Eastern Cooperative Oncology Group (ECOG) PS <2 (Appendix B).
* Previous treatment: Patients must have responded to first or second line hormonal therapy (Partial and complete response greater than 6 months using RECIST criteria. Patients with stable disease for more than 6 months will be eligible) and became resistant to the hormonal agent. They must remain on the current hormone therapy to which they initially responded but now are resistant.
* Clear documentation of acquired hormonal resistance.
* Evaluable disease will be considered eligible, but measurable disease according to RECIST criteria will be preferable (Appendix C). The target lesion(s) must not have been previously irradiated (newly arising lesions in previously irradiated areas are acceptable).
* Patients must have adequate organ and marrow function as defined as follows: absolute neutrophil count > 1,500/mm3, hemoglobin > 8.0 g/dl, platelets > 75,000/mm3, total bilirubin < 2 mg/dl, serum creatinine < 2 mg/dl, transaminases (AST, ALT) may be up to 2.5 x institutional upper limit of normal for patients with no liver metastases and up to 5 x institutional upper normal limit for patients with documented liver metastases. In addition < 1 gr of protein in 24 hr urine collection and urine protein/creatinine ratio < 1.0
* Prior chemotherapy does not exclude patients from study as long as the current therapy was hormonal therapy alone.
* Patients with de novo hormone therapy resistance will not be eligible.
* No life threatening parenchymal disease or rapidly progressing disease warranting cytotoxic chemotherapy.
* No history of brain metastases.
* No history of thrombosis during the previous year, including transient ischemic attack.
* Hypertension must be controlled (< 150/100 mmHg).
* Ejection Fraction > 50%.

Exclusion Criteria:

* Patients who are "de novo" resistant to hormone therapy.
* Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study other than this Genentech-sponsored bevacizumab cancer study.
* Blood pressure of >150/100 mmHg
* Unstable angina
* New York Heart Association (NYHA) Grade II or greater congestive heart failure
* History of myocardial infarction within 6 months
* History of stroke within 6 months
* Clinically significant peripheral vascular disease
* History of a bleeding disorder
* Presence of central nervous system or brain metastases
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0, anticipation of need for major surgical procedure during the course of the study
* Minor surgical procedures, fine needle aspirations or core biopsies within 7 days prior to Day 0
* Pregnant (positive pregnancy test) or lactating
* Urine protein: creatinine ratio greater than or equal to 1.0 at screening. Patients demonstrating > 1 gr of protein in 24 hr urine collection within 4 weeks prior to study entry will not participate in the trial.
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to Day 0
* Serious, non-healing wound, ulcer, or bone fracture
* Unwilling or unable to comply with the protocol for the duration of the study.
* Psychiatric illness/social situations that would limit compliance with study requirements.
* Previously radiated area(s) must not be the only site of disease.
* History of another malignancy within the last five years except cured basal cell carcinoma of skin and carcinoma in-situ of uterine cervix.

Ages: 19 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-10; Primary Completion 2009-03 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carla Falkson, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started October 2005 - until March 2009. Kirklin Clinic at University of Alabama at Birmingham (UAB), Birmingham, Alabama (AL) and Georgia Cancer Center, Atlanta, Georgia (GA)
Pre-assignment Details: The purpose of this study is to determine if acquired hormone therapy resistance can be reversed by Avastin (Bevacizumab), as measured by time to disease progression and evaluate toxicity of the combination of hormone treatment plus Avastin.
Groups:
- Avastin(Bevacizumab) Plus Hormonal Therapy: Avastin (Bevacizumab)15mg/m2 IV every 3 weeks plus various daily oral hormonal therapies.
Period: Overall Study
Arm/Group | Avastin(Bevacizumab) Plus Hormonal Therapy
Started | 30
Completed | 27 (3 patients withdrew consent after 29, 5 and 3 1/2 months on study.)
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Avastin(Bevacizumab) Plus Hormonal Therapy
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Progression free survival is defined as time from date of registration until the date of first documented disease progression or date of death from any cause, whichever occurs first.
Time Frame: From date of registration until disease progression or death, whichever occurs first
Population: All participants entered onto study (intention to treat) (ITT) were analyzed.
Measure: Median (95% Confidence Interval); unit: days
Groups:
- Avastin (Bevacizumab) Plus Hormone: All patients received Avastin (Bevacizumab) 15 mg/kg IV every three weeks as well as continuing with hormonal therapy they previously were taking.
Arm/Group | Avastin (Bevacizumab) Plus Hormone
Number analyzed (Participants) | 30
days | 125.5 [90 to 256]

2. Secondary Outcome: Objective Response Rate (Defined as the Rate of Complete and Partial Responses).
Time Frame: From date of registration until disease progression or death, whichever occurs first
Measure: Number; unit: participants
Arm/Group | Avastin
Number analyzed (Participants) | 30
participants | 0

ADVERSE EVENTS:
Time Frame: 1245 days
Arm/Group | Avastin(Bevacizumab) Plus Hormonal Therapy
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 7/30
Other Adverse Events (participants affected / at risk) | 24/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Avastin(Bevacizumab) Plus Hormonal Therapy (N=30)
Grade III diarrhea (Gastrointestinal disorders) | 1
Grade III leg ulcer (Skin and subcutaneous tissue disorders) | 1
Grade III fatigue (General disorders) | 2
Grade III hypertension (Vascular disorders) | 4
Grade III neuropathy (Nervous system disorders) | 1
Grade III syncope (General disorders) | 2
Knee and foot pain (Musculoskeletal and connective tissue disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Grade III dyspnea on exertion (Respiratory, thoracic and mediastinal disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Avastin(Bevacizumab) Plus Hormonal Therapy (N=30)
Proteinuria (Renal and urinary disorders) | 10
Diarrhea (Gastrointestinal disorders) | 3
Hoarsness of voice (Respiratory, thoracic and mediastinal disorders) | 3
Transaminitits (Gastrointestinal disorders) | 4
Fatigue (General disorders) | 6
Hypertension (Vascular disorders) | 4
Nausea and vomiting (Gastrointestinal disorders) | 8
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Ear and labyrinth disorders) | 4
GI Bleeding (Gastrointestinal disorders) | 2
Acute Renal Failure (Renal and urinary disorders) | 2
Dizziness (Ear and labyrinth disorders) | 2
Anorexia (General disorders) | 2
Weight loss (General disorders) | 4
Anemia (Blood and lymphatic system disorders) | 2
Mucositis (Gastrointestinal disorders) | 4
Change in taste (Gastrointestinal disorders) | 2
Skin rash (Skin and subcutaneous tissue disorders) | 2
Headache (Nervous system disorders) | 2
Arthralgias (Musculoskeletal and connective tissue disorders) | 2

LIMITATIONS AND CAVEATS:
A Phase II trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No